CLINICAL TRIAL: NCT04298515
Title: Determination of the Relationship Between Nesfatin-1 Levels and Energy Intake Levels of Patients With Type 2 Diabetes, Insulin Resistance and Obesity
Brief Title: Nesfatin-1 Level in Patients With Type 2 Diabetes, Insulin Resistance and Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Gülin Öztürk Özkan, Assistant Professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: HNEAH-KAEK 2019/100
Record Dates: First submitted 2020-02-10; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes; Insulin Resistance; Obesity; Nesfatin-1
Keywords: Type 2 diabetes; Insulin resistance; Obesity; Nesfatin-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Type 2 Diabetes group (Other): In case of fasting, blood will be taken from patients for the measurement of nesfatin-1.
  Interventions: Diagnostic Test: Nesfatin-1
- Insulin resistance group (Other): In case of fasting, blood will be taken from patients for the measurement of nesfatin-1.
  Interventions: Diagnostic Test: Nesfatin-1
- Obesity group (Other): In case of fasting, blood will be taken from patients for the measurement of nesfatin-1.
  Interventions: Diagnostic Test: Nesfatin-1

INTERVENTIONS:
Diagnostic Test: Nesfatin-1 — Blood will be taken from the patients on an empty stomach for measuring nesfatin-1 level

SUMMARY:
This research was planned to determine the level of nesfatin-1, known as satiety hormone, in type 2 diabetes, insulin diabetes and obesity patients and to determine whether there is a relationship between patients' energy intake levels. Additionally, it was aimed to evaluate the relationship between patients' nesfatin-1 values and serum glucose, insulin, lipid concentrations.

DETAILED DESCRIPTION:
Nesfatin-1 levels of patients with type 2 diabetes, insulin resistance and obesity will be measured. In addition, patients' daily food consumption will be taken and the amount of energy they receive will be calculated daily. The relationship between the level of nesfatin-1 in the blood and the energy received will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Insulin resistance
* Obesity disease

Exclusion Criteria:

* Pediatric individuals
* All patients who are hospitalized,
* Liver disease
* Cancer patients
* Disease related to the gastrointestinal tract
* Nephrological disease such as chronic kidney failure, acute kidney failure, nephrotic syndrome
* Neurological disease

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-03-02 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Nefratin-1 in type 2 diabetes | 1 day (Blood will be drawn from patients once)
  Blood will be drawn from type 2 diabates patients after 12 hours of fasting (n=45)
Nefratin-1 in obesity | 1 day (Blood will be drawn from patients once)
  Blood will be drawn from obesity patients after 12 hours of fasting (n=45)
Nefratin-1 in insulin resistance | 1 day (Blood will be drawn from patients once)
  Blood will be drawn from insulin resistance patients after 12 hours of fasting (n=45)

CONTACTS AND LOCATIONS:
Overall Officials: Gülin Öztürk Özkan, Assis Prof, Study Chair — İstanbul Medeniyet University; Kadir Kayataş, associate professor, Study Director — Haydarpaşa Numune Education and Research Hospital
Locations (1):
- Haydarpaşa Numune Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dore R, Levata L, Lehnert H, Schulz C. Nesfatin-1: functions and physiology of a novel regulatory peptide. J Endocrinol. 2017 Jan;232(1):R45-R65. doi: 10.1530/JOE-16-0361. Epub 2016 Oct 17. PMID 27754932
- [Background] Mirzaei K, Hossein-nezhad A, Keshavarz SA, Koohdani F, Eshraghian MR, Saboor-Yaraghi AA, Hosseini S, Chamari M, Zareei M, Djalali M. Association of nesfatin-1 level with body composition, dietary intake and resting metabolic rate in obese and morbid obese subjects. Diabetes Metab Syndr. 2015 Oct-Dec;9(4):292-8. doi: 10.1016/j.dsx.2014.04.010. Epub 2014 May 25. PMID 25470645
- [Result] Li QC, Wang HY, Chen X, Guan HZ, Jiang ZY. Fasting plasma levels of nesfatin-1 in patients with type 1 and type 2 diabetes mellitus and the nutrient-related fluctuation of nesfatin-1 level in normal humans. Regul Pept. 2010 Jan 8;159(1-3):72-7. doi: 10.1016/j.regpep.2009.11.003. PMID 19896982
- See also: Review — http://www.ncbi.nlm.nih.gov/pubmed/?term=10.1530%2FJOE-16-0361
- See also: Original research — http://www.ncbi.nlm.nih.gov/pubmed/?term=19896982
- See also: Original research — http://www.ncbi.nlm.nih.gov/pubmed/?term=10.1016%2Fj.dsx.2014.04.010